CLINICAL TRIAL: NCT04600128
Title: The Effect of Pre-meal Serving of Dairy and Dairy Alternatives on Post-meal Satiety, Food Intake, and Glycaemia in Healthy Young Adults
Brief Title: Effect of Pre-meal Serving of Dairy and Dairy Alternatives on Post-meal Satiety and Glycaemia in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DFC_31323_PlantProtein
Record Dates: First submitted 2020-10-21; First posted 2020-10-23 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Dairy; Yogurt; Cheese; Postprandial glycaemia; Satiety; Plant based dairy alternative
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dairy-based Greek yogurt (Active Comparator): Plain dairy-based Greek yogurt
  Interventions: Other: Dairy-based greek yogurt
- Dairy-based cheddar cheese (Active Comparator): Mild dairy-based cheddar cheese
  Interventions: Other: Dairy-based cheddar cheese
- Plant-based Greek yogurt (Active Comparator): Plain plant-based Greek yogurt
  Interventions: Other: Plant-based yogurt
- Plant-based cheese (Active Comparator): Medium cheddar plant-based cheese
  Interventions: Other: Plant-based cheese

INTERVENTIONS:
Other: Dairy-based greek yogurt — Plain Greek yogurt (2% M.F; Danone, Boucherville, Quebec, Canada)
  Arms: Dairy-based Greek yogurt
Other: Dairy-based cheddar cheese — Mild cheddar cheese (31% M.F. ; Armstrong, Saputo Dairy Products, Saint-Laurent, Quebec, Canada)
  Arms: Dairy-based cheddar cheese
Other: Plant-based yogurt — Plain Greek yogurt alternative (Daiya, Rupert Street, Vancouver, Canada)
  Arms: Plant-based Greek yogurt
Other: Plant-based cheese — Medium cheddar style block (Daiya, Rupert Street, Vancouver, Canada)
  Arms: Plant-based cheese

SUMMARY:
Regular consumption of dairy products is found to negatively associated with metabolic diseases and improve body composition in long term studies and has positive effect on acute glycemia control and satiety. However, new Canada's Food Guide released in 2019 promotes a shift from traditional dairy products to plant-based dairy alternatives. The present study examines the effect of traditional dairy products in comparison with plant-based alternatives on glycemic response and satiety.

DETAILED DESCRIPTION:
In the past forty years, the prevalence of obesity in adults has doubled, and nearly two thirds of Canadian adults are currently overweight or obese (Kenneth and Eggleton,2016). The incidence of diabetes, heart disease, stroke and certain cancers has also increased correspondingly (Xavier P. 2010). Obesity not only leads to other chronic diseases but also decreases life expectancy and puts a strain on the health care system (Tremmel 2017). Therefore, it is important to find strategies to minimize obesity and type-2 diabetes. Postprandial glycemia (PPG) has been identified to be one of the implications of risk factor of metabolic diseases such as obesity (Black 2012). To better help identify foods that increase satiety and decrease PPG, Health Canada released a draft guidance document to validate health food claims related to "reduction of post-prandial glycaemic response" (Health Canada 2013).

Regular consumption of dairy products correlates with improved body composition and lower incidences of obesity and type 2 diabetes in both observational and long-term clinical studies (Hirahatake et al. 2014; Lee et al. 2018; Murphy et al. 2013; Soedamah-Muthu and de Goede 2018). Within typical dietary patterns, high-fat dairy consumption is inversely associated with the risk of obesity or overweight (Kratz et al. 2013; Rautiainen et al. 2016). Frequent cheese consumption was associated with lower BMI in a 10 year follow-up study (Guo et al. 2018). The hypothesis that these associations between dairy and obesity and chronic metabolic diseases can be attributed to lasting metabolic effects of dairy when consumed with high glycemic carbohydrate or as a between meal snack is supported by short term studies. A recent meta-analysis of clinical trials concluded that, dairy products when consumed alone result in significant decreases in appetite and later energy intake (Onvani et al. 2017). Other recent studies have shown that milk consumed with a high glyemic breakfast cereal significantly reduced PPG as well as appetite in both young (Kung et al. 2018; Law et al. 2017a) and older adults (Law et al. 2017b). Among dairy products, semi solid and solid dairy products such as cheese and yogurt consumed with carbohydrates increased satiety and lowered PPG more than milk or soy beverages (Law et al. 2017b). PPG and appetite were significantly reduced following single serving amounts, of skim-milk, full fat milk, yogurt and cheese when consumed alone (Vien et al. 2019). Appetite measured over three hours was reduced after dairy consumption compared to a water control, particularly skim milk reducing appetite more than full fat milk, yogurt or cheese. Over 120 minutes, PPG was the lowest after cheese (Vien et al. 2019).

This data suggests that dairy consumed immediately before a meal will affect satiety and glycemic responses to a later meal, but the response will depend on the type of dairy product consumed. The updated Canada's Food Guide promotes the consumption of plant-based protein and a shift away from consuming dairy products as plant-based products may provide more fibre and less saturated fat (Canada Food Guide 2019). As a result, many plant based dairy substitutes have appeared in the marketplace. However, these new products, in addition to being of low protein quality, my lack the physiological functionality of dairy in metabolic regulation.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18.5-24.9 kg/m^2

Exclusion Criteria:

* smoke
* skip breakfast
* lactose intolerant
* allergic to study foods
* dislike study foods
* are not comfortable with finger pricking
* take prescription medication less than a year
* undergoing hormonal treatments for less than 1 year
* trying to gain or lose weight
* have diabetes or cardiovascular disease
* restrained eaters (identified by a score of ≥ 11 using the Eating Habits Questionnaire)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose levels | Starting at the beginning of each session (0 minutes before consumption of treatment) and every 15-30 minutes up to 160 minutes (time of completion of each session)
  Blood glucose (mmol/L) is measured using finger prick capillary blood samples

OTHER OUTCOMES:
Subjective appetite | up to 160 minutes (time of completion of each session)
  Measured using Visual Analog Scales (VAS). Subjective appetite is determine by desire to eat, hunger, fullness, and prospective consumption. The scale is 0 to 100 where zero indicates low desire to eat, hunger, prospective consumption and lesser fullness. One hundred indicates high desire to eat, hunger, prospective consumption, and greater fullness,
Insulin | up to 160 minutes (time of completion of each session)
  Blood insulin (μU/mL) is measured using finger prick capillary blood samples

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Da Silva N, Anderson G, Amr A, Vien S, Fabek H. A comparison of the effects of dairy products with their plant-based alternatives on metabolic responses in healthy young Canadian adults: a randomized crossover study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-17. doi: 10.1139/apnm-2024-0158. PMID 39146559